CLINICAL TRIAL: NCT01027780
Title: Mindfulness to Improve Elders' Immune and Health Status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Jan Moynihan, Director, The Rochester Center for Mind-Body Research, University of Rochester Medical Center, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R01AG025474 (NIH); R01AG025474 (NIH)
Record Dates: First submitted 2009-12-06; First posted 2009-12-09 (Estimated); Results first posted 2014-08-27 (Estimated); Last update posted 2014-08-27 (Estimated); Status verified 2014-01

CONDITIONS: Stress, Psychologic
Keywords: Mindfulness-Based Stress Reduction; MBSR; Seniors; immune system; keyhole limpet hemocyanin (KLH)
MeSH Terms: conditions — Stress, Psychological | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mindfulness-Based Stress Reduction (Active Comparator): Participation in the Mindfulness-Based Stress Reduction (MBSR) program following the initial assessment period, just prior to the start of the immunological measures.
  Interventions: Behavioral: Mindfulness-Based Stress Reduction
- Wait-list control (No Intervention): Wait-list control participants were offered MBSR training after completion of their primary assessments periods.

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction — The standardized Mindfulness-Based Stress Reduction (MBSR) program is the primary training tool used to enhance mindfulness. The eight-week-long MBSR program is designed to teach subjects how to develop their inner resources in the service of taking better care of themselves. MBSR training includes the learning and refining of a range of skills aimed at increasing relaxation and awareness of physical experiences and sensations related to physical symptoms, emotions, and thoughts. Special emphasis is placed on movement, meditation, and breathing.
  Other Names: MBSR
  Arms: Mindfulness-Based Stress Reduction

SUMMARY:
The purpose of the study is to better understand effects of the Mindfulness-Based Stress-Reduction (MBSR) program on the physical and emotional health and well-being of adults ages 65 and older.

The effects MBSR may have on the immune system is investigated, including how these effects relate to factors such as perceived health, psychological well-being, age, personality, and mood.

DETAILED DESCRIPTION:
This study investigates the effects of Mindfulness-Based Stress Reduction (MBSR) on immune responses to multiple concentrations of keyhole limpet hemocyanin (KLH) in elderly volunteers. The research design thus capitalizes on the antibody response to a novel, benign antigen to which our subjects will be immunologically naïve. The use of a range of antigen concentrations will provide a sensitive indicator for the effects of intervention.

The Aims of the study are the following:

1. To examine the effects of Mindfulness Based Stress Reduction (MBSR) on immunological outcomes, perceived health, and psychological well-being in a sample of seniors 65 years of age and older.
2. To examine whether treatment effects are moderated by age, personality traits, physical health status, or depression.
3. To examine the effects of behavioral, psychological, and physiological mediators of immune outcome.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 or older
* English speaking
* If prescribed antidepressant or anxiolytic medications, must have maintained a stable regimen for eight weeks prior to enrolling

Exclusion Criteria:

* receiving immunosuppressive therapy for cancer or other diseases
* major, uncorrected sensory impairments
* cognitive deficits (MMSE <25, or deficits deemed significant enough to interfere)
* history of a psychotic disorder, bipolar disorder, organic brain syndrome, or mental retardation
* alcohol or substance abuse within the previous year
* severe cardiovascular disease
* known allergies to shellfish

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 208 (Actual)
Dates: Start 2006-03; Primary Completion 2009-05 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan A Moynihan, Ph.D, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

REFERENCES:
- [Result] Gallegos AM, Hoerger M, Talbot NL, Moynihan JA, Duberstein PR. Emotional benefits of mindfulness-based stress reduction in older adults: the moderating roles of age and depressive symptom severity. Aging Ment Health. 2013;17(7):823-9. doi: 10.1080/13607863.2013.799118. Epub 2013 May 22. PMID 23697871
- [Result] Gallegos AM, Hoerger M, Talbot NL, Krasner MS, Knight JM, Moynihan JA, Duberstein PR. Toward identifying the effects of the specific components of Mindfulness-Based Stress Reduction on biologic and emotional outcomes among older adults. J Altern Complement Med. 2013 Oct;19(10):787-92. doi: 10.1089/acm.2012.0028. Epub 2013 Feb 5. PMID 23383976
- [Result] Moynihan JA, Chapman BP, Klorman R, Krasner MS, Duberstein PR, Brown KW, Talbot NL. Mindfulness-based stress reduction for older adults: effects on executive function, frontal alpha asymmetry and immune function. Neuropsychobiology. 2013;68(1):34-43. doi: 10.1159/000350949. Epub 2013 Jun 15. PMID 23774986
- [Result] Chapman BP, van Wijngaarden E, Seplaki CL, Talbot N, Duberstein P, Moynihan J. Openness and conscientiousness predict 34-week patterns of Interleukin-6 in older persons. Brain Behav Immun. 2011 May;25(4):667-73. doi: 10.1016/j.bbi.2011.01.003. Epub 2011 Jan 15. PMID 21241793
- [Derived] Gallegos AM, Moynihan J, Pigeon WR. A Secondary Analysis of Sleep Quality Changes in Older Adults From a Randomized Trial of an MBSR Program. J Appl Gerontol. 2018 Nov;37(11):1327-1343. doi: 10.1177/0733464816663553. Epub 2016 Aug 10. PMID 27511921

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between March 2006 and August 2009, women and men ages 65 and older were recruited from the community via advertisements in local newspapers and from University of Rochester Strong Health-associated primary care offices using flyers. Exclusion criteria were utilized as indicated in the protocol section.
Period: Overall Study
Arm/Group | Mindfulness-Based Stress Reduction | Wait-list Control
Started | 105 | 103
Completed | 105 | 102
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindfulness-Based Stress Reduction | Wait-list Control | Total
Number analyzed (Participants) | 105 | 103 | 208
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 103 | 102 | 205
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.3 (6.7) | 73.6 (6.7) | 73.02 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 64 | 129
  Male | 40 | 39 | 79
Region of Enrollment [Number; unit: participants]
  United States | 105 | 103 | 208

OUTCOME MEASURES:

1. Primary Outcome: IgG Anti-KLH Antibody Response Post-treatment
Description: Immune function--specifically, antibody response to a novel, benign antigen (an antigen to which subjects are immunologically naïve); in this case, keyhole limpet hemocyanin (KLH).
Time Frame: Immediate post-treatment (time 2)
Measure: Mean (Standard Error); unit: OD 405 nm
Arm/Group | Mindfulness-Based Stress Reduction | Wait-list Control
Number analyzed (Participants) | 105 | 103
OD 405 nm | 0.172 (.04) | 0.104 (.032)
Statistical Analysis 1: Comparison: Mindfulness-Based Stress Reduction vs Wait-list Control; Test type: Superiority or Other; p = .007, GEE — Please note that this analysis tested the differences between groups following the intervention; Generalized estimating equations (GEE) approach was used to assess robustness of population parameters, such as treatment effects

2. Primary Outcome: Trail Making Test
Description: The Trail Making Test is a commonly used neuropsychological test of visual attention and task-switching. In two timed tasks, subjects are asked to first connect numbers (Test A), then alternating numbers and letters (Test B), in sequential order as quickly as possible. Completion times, relating to cognitive processing speed and executive function (respectively), may be utilized individually, and as a difference (B-A) or ratio (B/A) score. The Trails B/A ratio was used as an index of improvement in executive control throughout the trial, with lower scores indicating better performance.
Time Frame: immediate post-treatment (Time 2)
Measure: Mean (Standard Error); unit: Trails B:A score
Arm/Group | Mindfulness-Based Stress Reduction | Wait-list Control
Number analyzed (Participants) | 105 | 103
Trails B:A score | 1.75 (.1) | 2.01 (.11)
Statistical Analysis 1: Comparison: Mindfulness-Based Stress Reduction vs Wait-list Control; Test type: Superiority or Other; p = .04, GEE — Note that this is the p value for differences between groups immediately following the intervention; [statistical method as in outcome 1, analysis 1]

3. Primary Outcome: Electroencephalography Measurement
Description: Measurement of alpha asymmetry at the F3/4 (frontal) electrode. Left prefrontal activation has been associated with positive affect, and with higher levels of antibody responses and natural killer cell cytotoxicity.
Time Frame: post-treatment (time 2)
Population: Some subject EEG recordings were excluded from analyses due to reading/equipment factors (e.g., poor signal, external noise) or subject factors (e.g., sleepiness, illness). Subjects were also allowed to opt out of the EEG procedures if desired.
Measure: Mean (Standard Error); unit: Log right-log left alpha power
Groups:
- Mindfulness Based Stress Reduction: Participation in the Mindfulness-Based Stress Reduction (MBSR) program following the initial assessment period, just prior to the start of the immunological measures.
Arm/Group | Mindfulness Based Stress Reduction | Wait-list Control
Number analyzed (Participants) | 55 | 55
Log right-log left alpha power | 0.067 (.03) | -0.25 (.03)
Statistical Analysis 1: Comparison: Mindfulness Based Stress Reduction vs Wait-list Control; Test type: Superiority or Other; p = .03, ANOVA — Difference between groups following intervention

ADVERSE EVENTS:
Arm/Group | Mindfulness-Based Stress Reduction | Wait-list Control
Serious Adverse Events (participants affected / at risk) | 0/105 | 0/103
Other Adverse Events (participants affected / at risk) | 0/105 | 0/103

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No